CLINICAL TRIAL: NCT07191002
Title: The Role of Existing Formulas and Airway Measurements in Determining the Appropriate Placement Depth of the Double-lumen Tube in Thoracic Surgery Anesthesia: a Prospective Observational Study
Brief Title: The Role of Existing Formulas in the Double-lumen Tube in Thoracic Surgery Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Baldemir, Clinic Associate Professor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2024-BÇEK/344
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Double-lumen Tube; One-lung Ventilation (OLV); Thoracic Anesthesia
Keywords: Double-Lumen Tube; Fiberoptic Bronchoscopy; Airway Measurements; One-Lung Ventilation; Tube Placement Depth; Thoracic Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intubated with a left DLT: Patients who will undergo surgery under general anesthesia and be intubated with a left DLT
  Interventions: Other: placement depth of the double lumen tube

INTERVENTIONS:
Other: placement depth of the double lumen tube — the anesthesiologist will select the appropriate DLT size and placement depth entirely at their discretion, as per routine practice, and confirm both using fiberoptic bronchoscopy (FOB). If malposition occurs, it will be corrected under FOB guidance, and the tube will be secured in the correct position

SUMMARY:
In most clinical scenarios, left DLT is preferred for one-lung ventilation because of its anatomical ease of placement; these tubes allow separate ventilation of both lungs. If the DLT is not placed in the proper size and depth, it may result in repeated intubation attempts, airway and dental trauma, failed lung isolation, tube dislodgement, and various unwanted events such as hypoxemia.

The first and most common method for correct placement of a DLT is the conventional technique, blindly advanced into the left main bronchus, and then confirmed with fiberoptic bronchoscopy (FOB). In this method, the depth at which the tube should be left before performing FOB is left to the clinician's experience. Generally, the DLT is advanced in the trachea until a slight resistance is felt. This may lead to excessive advancement of the DLT into the left main bronchus or premature resistance due to the tube tip touching the carina, causing the clinician to stop before entering the left main bronchus. Therefore, just as selecting the correct size of the DLT is crucial, correctly estimating the appropriate depth is also of great importance. For this reason, different formulas have been proposed in the literature, and new formulas are still being investigated.

The patient's gender and height are determinant in selecting the appropriate size of the DLT. However, studies in the literature indicate that the accuracy of these formulas may be limited in Asian populations. Therefore, it is important to evaluate the applicability of these formulas in different populations and, if necessary, develop new formulas. In the Turkish population as well, verifying the accuracy of these formulas for determining the proper size and depth of DLT-and if needed, developing new recommendations and formulas-holds clinical importance.

In this study, conducted at Ankara Atatürk Sanatorium Training and Research Hospital, the aim is to evaluate the accuracy of six different formulas available in the literature for predicting DLT depth in patients undergoing thoracic surgery. Additionally, the correlations between DLT depth and demographic parameters as well as external airway measurements (mouth opening, sternomental distance, thyromental distance, distance between the mentum and manubrio-sternal angle, distance between tragus and manubrio-sternal angle, distance between sternal angle and xiphoid process) will be analyzed. Furthermore, challenges during DLT application, malposition rates and types, and complications will be assessed.

The primary objective of this study is to evaluate, in patients undergoing thoracic surgery at Ankara Atatürk Sanatorium Training and Research Hospital, how accurate and applicable six different formulas defined in the literature are for predicting the placement depth of the DLT. If the existing formulas are insufficient, the aim is to develop a new formula.

DETAILED DESCRIPTION:
Hypothesis H0 (Null Hypothesis): The formulas defined in the literature accurately predict the placement depth of the left double-lumen tube (DLT) in the Turkish population; therefore, no additional measurement methods are required.

H1 (Alternative Hypothesis): The formulas defined in the literature do not accurately predict the placement depth of the left double-lumen tube (DLT) in the Turkish population; therefore, DLT placement depth can be predicted more accurately using external anatomical parameters and population-specific measurement methods, and additional measurement methods are required.

Study Design The study has been designed as a single-center, prospective observational study.

Study Setting/ Location The study will be conducted at Ankara Atatürk Sanatorium Training and Research Hospital, in the Department of Anesthesiology and Reanimation, Thoracic Surgery operating room.

Study Population The study will begin prospectively after obtaining approval from the ethics committee and will be completed once the target number of patients has been reached. The study population will consist of patients aged 18-80 years who will undergo thoracic surgery at the operating rooms of the Department of Anesthesiology and Reanimation, Ankara Atatürk Sanatorium Training and Research Hospital.

Inclusion Criteria:

* Patients older than 18 and younger than 80 years
* Patients who will undergo surgery under general anesthesia and be intubated with a left DLT
* Patients with an American Society of Anesthesiologists (ASA) score of I-II-III
* Patients with a body mass index (BMI) between 18-40 kg/m²
* Patients who provide informed consent

Exclusion Criteria:

* Patients requiring right DLT placement
* Patients with ASA score IV and above
* Patients intubated with a single-lumen tube
* Patients in whom lung isolation will be achieved with a method other than DLT
* Emergency cases
* Patients younger than 18 or older than 80 years Primary and Secondary Outcome

Primary Outcome:

The primary outcome of the study is the consistency between the DLT depths calculated using six different formulas defined in the literature and the actual placement depth confirmed by fiberoptic bronchoscopy (FOB).

Secondary Outcomes:

1. The relationship between external anatomical measurements (mouth opening, sternomental distance, thyromental distance, distance between mentum and manubrio-sternal angle, distance between tragus and manubrio-sternal angle, distance between sternal angle and xiphoid process) and DLT depth.
2. The correlation between patients' demographic characteristics (height, weight, sex, body mass index) and DLT placement depth.
3. The frequency of technical difficulties encountered during DLT placement (e.g., difficulty in intubation, intubation time, need for maneuvers, requirement for repositioning).
4. Distribution of malposition rates and types (early, late; proximal and distal positioning, etc.).
5. Frequency and types of complications (e.g., hypoxemia, airway trauma, dental injury, tube dislodgement, etc.).
6. If existing formulas are found to be inconsistent, development of a new formula specifically for the Turkish population.

This thesis study will be conducted in accordance with the Declaration of Helsinki and, after obtaining approval from the relevant units and the ethics committee, will be carried out at Ankara Atatürk Sanatorium Training and Research Hospital.

Patients aged 18-80 years who will undergo thoracic surgery and agree to participate in the study by signing the informed consent form will be prospectively enrolled. A total of 30 patients will be included in the study. All patients will be informed about the study process, and informed consent will be obtained.

Inclusion criteria: patients over 18 and under 80 years of age, intubated with a left DLT, American Society of Anesthesiologists (ASA) score I-II-III, body mass index (BMI) between 18-40 kg/m², and undergoing surgery under general anesthesia.

Exclusion criteria: patients requiring right DLT placement, patients with ASA IV and above, patients intubated with a single-lumen tube, patients in whom lung isolation is achieved by a method other than DLT.

During routine preoperative anesthesia evaluation, demographic data such as age, height, body weight, body mass index (BMI), sex, comorbidities, prior surgeries, ASA score, Mallampati classification, mouth opening, sternomental distance, thyromental distance, distance between mentum and manubrio-sternal angle, distance between tragus and manubrio-sternal angle, and distance between sternal angle and xiphoid process will be recorded.

No additional procedures specific to this study will be performed. After anesthesia induction, the anesthesiologist will select the appropriate DLT size and placement depth entirely at their discretion, as per routine practice, and confirm both using fiberoptic bronchoscopy (FOB). If malposition occurs, it will be corrected under FOB guidance, and the tube will be secured in the correct position. No intervention or guidance will be given to the anesthesiologist during this process.

After DLT placement, the insertion depth will be measured at the corner of the mouth. During DLT application, any difficulties encountered, malposition rates and types, complications, and perioperative or postoperative events related to DLT use (such as hoarseness, sore throat, dental injury, lip or oral trauma, cough) will be recorded. Hemodynamic parameters (systolic arterial pressure [SAP], diastolic arterial pressure [DAP], mean arterial pressure [MAP], heart rate, oxygen saturation) will be recorded at the following time points: before induction, after induction, immediately after intubation, just before extubation, and immediately after extubation.

The study is planned to be completed within 3-6 months after obtaining ethics committee approval. It will be terminated once the target study population is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and younger than 80 years
* Patients who will undergo surgery under general anesthesia and be intubated with a left DLT
* Patients with an American Society of Anesthesiologists (ASA) score of I-II-III
* Patients with a body mass index (BMI) between 18-40 kg/m²
* Patients who provide informed consent

Exclusion Criteria:

* Patients requiring right DLT placement
* Patients with ASA score IV and above
* Patients intubated with a single-lumen tube
* Patients in whom lung isolation will be achieved with a method other than DLT
* Emergency cases
* Patients younger than 18 or older than 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will begin prospectively after obtaining approval from the ethics committee and will be completed once the target number of patients has been reached. The study population will consist of patients aged 18-80 years who will undergo thoracic surgery at the operating rooms of the Department of Anesthesiology and Reanimation, Ankara Atatürk Sanatorium Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
consistency between the DLT depths calculated using six different formulas | during perioperative
  The primary outcome of the study is the consistency between the DLT depths calculated using six different formulas defined in the literature and the actual placement depth confirmed by fiberoptic bronchoscopy (FOB).

CONTACTS AND LOCATIONS:
Overall Officials: ELİF DURMUŞ, Principal Investigator — ANKARA ATATURK SANATORİUM TRAİNİNG AND RESEARCH HOSPITAL
Locations (1):
- Ankara Ataturk Sanatorium Training and Research Hospital, Ankara, 06280, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No